CLINICAL TRIAL: NCT00001244
Title: Studies of Immune Regulation in Patients With Common Variable Immunodeficiency and Related Inborn Errors of Immunity (IEI)
Brief Title: Immune Regulation in Patients With Common Variable Immunodeficiency and Related Inborn Errors of Immunity (IEI)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890158; 89-I-0158
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-05-13

CONDITIONS: XLA; CVID; Yao Syndrome; Blau Syndrome
Keywords: Blau Syndrome; XLA; Humoral Immunodeficiency; CVID enteropathy; CVID; Agammaglobulinemia; Inborn Errors of Immunity; Yao Syndrome
MeSH Terms: conditions — Blau syndrome; Agammaglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Population: Physician referral required

SUMMARY:
This study aims to understand the causes and progression of Common Variable Immunodeficiency (CVID) and related inborn errors of immunity (IEI). These are conditions where the immune system does not function properly, leading to frequent infections and other complications such as gastrointestinal inflammation, lung and liver disease, autoimmune conditions, and an increased risk of certain cancers. By studying patients with CVI and related immune disorders, we hope to develop better ways to diagnose, treat, and prevent complications associated with these conditions.

Patients diagnosed with CVID or related immune disorders must be referred by their physician and medical records reviewed by the study team to confirm eligibility to participate in this study. Once enrolled, participants will undergo various tests, including blood draws, physical exams, and imaging studies like CT scans to track changes over time. We may collect samples such as blood, urine, stool, or saliva for research purposes. If a surgical procedure or biopsy is performed because it is medically necessary, we may collect an additional sample for research testing. Family members of patients may be asked to provide blood samples for comparison. Some tests may be done remotely if participants or family members cannot travel to the study site.

Who Can Participate

* Patients diagnosed with CVI or related IEI, such as X-linked agammaglobulinemia, Blau Syndrome or Yao Syndrome.
* Participants must be at least 2 years old.
* Family members of patients may include parents, siblings, grandparents, children, aunts, uncles, and cousins.
* Pregnant women already enrolled in the study will continue to participate, but new pregnant participants will not be enrolled.

Potential Risks and Benefits

* Risks: Blood draws may cause discomfort, bruising, or infection. Apheresis may cause dizziness, nausea, or muscle cramps; this procedure is to collect specific cells in the blood and is infrequently done on this protocol. Extra biopsies during clinically indicated procedures may increase the risk of complications; they will only be collected after the medically necessary biopsies are taken and if it is safe to collect any extra biopsies.
* Benefits: Participants may not receive direct medical benefits, but the study will contribute to a better understanding of CVID and related conditions, potentially leading to improved treatments.

DETAILED DESCRIPTION:
The purpose of this protocol is to carry out laboratory studies concerning the immunopathogenesis of Common Variable Immunodeficiency (CVI) and related inborn errors of immunity (IEI). Additionally, we aim to document and track the progression of known complications of these immune abnormalities. Complications associated with CVI include recurrent respiratory, granulomas, pulmonary insufficiency, gastrointestinal bacterial infections, enteropathy, nodular regenerative hyperplasia, lymphoid malignancy, and various autoimmune manifestations.

Patients with CVI and related IEI will be enrolled into this natural history study. Protocol procedures will include baseline measurements of and changes in lab studies. First- or second-degree genetically related family members (limited to mother, father, siblings, grandparents, children, aunts, uncles, and first cousins of an affected patient) may also be screened for clinical, in vitro, and genetic correlates of immune abnormalities. Changes in the patients' clinical state will be measured to determine the precursors of disease complications. This may lead to developments in improving preventive measures and novel treatment options for this population.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have a verifiable diagnosis of common variable immune deficiency as defined by a decrease both in IgG and at least one other Ig isotype to below two standard deviations of normal control levels OR B-cell immunodeficiencies related to CVI (defined as selective IgA deficiency, selective IgG isotype deficiency, agammaglobulinemia, and hypogammaglobulinemia associated with Epstein-Barr virus infection), or hypogammaglobulinemia associated with other related inborn errors of immunity. This includes patients with a defined diagnosis of Blau or Yao Syndrome.
* Must be 2 years old or greater.
* Patients with repeated infections and suspected of having an inborn error of immunity.
* Patients must be referred by their primary medical care provider.
* On investigator s discretion, unaffected family members (mother, father, siblings, children, grandparents, aunts, uncles, and first cousins) may be asked for the provision of blood or buccal specimens for research purposes.
* Patients who are lactating, may be eligible and will only undergo tests and procedures, and/or receive medications for which data exists that proves that they are minimal risk to the child.
* Pregnant women will not be newly enrolled onto this protocol, however existing patients who become pregnant while on study will remain on study, as literature about pregnancy in CVI patients is sparse and outside providers have minimal knowledge about managing CVI during pregnancy. Pregnant women will only undergo tests and procedures, and/or receive medications for which data exists that proves that they are minimal risk to the fetus. Pregnant unaffected relatives will not be enrolled in this study).
* All patients must be willing to have research samples stored for future studies and/or other research purposes.
* NIH staff and family members of study team members may be enrolled in this study as this population may meet study criteria. Neither participation nor refusal to participate as a subject in the research will have an effect, either beneficial or adverse, on the participant s employment or position at the NIH. Every effort will be made to protect participant information, but such information may be available in medical records and may be available to authorized users outside of the study team in both an identifiable and unidentifiable manner. The NIH investigator will provide and request that the NIH staff member review the Frequently Asked Questions (FAQs) for Staff Who are Considering Participating in NIH Research and the Leavy Policy for NIH Employees Participating in NIH Medical Research Studies (NIH Policy Manual 2300-630-3).

EXCLUSION CRITERIA:

* Presence of other medical illnesses that would preclude individuals from undergoing routine diagnostic testing or testing for immunologic features of immunodeficiency.
* Presence of a condition or treatment, such as HIV, cytotoxic chemotherapy or malignancy, that in the investigator s opinion could interfere with evaluation of the condition under study.
* Pregnancy at the time of enrollment.
* Inability of an adult participant to provide informed consent for themselves (decisionally impaired adult).

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population - Physician referral required
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1990-01-15 (Actual)

PRIMARY OUTCOMES:
Establish pattern/pace of disease process | At 1 year and ongoing
  To establish the pattern and pace of change of disease (frequency, distribution, type and extent of infections, inflammatory lesions and abnormalities of immune function).
Evaluation of organ dysfunction/damage resulting from immune abnormality | Ongoing
  To establish the extent of organ involvement (infection and/or inflammation) and organ damage or dysfunction resulting from the abnormality of immune function.
Characterization of immune abnormalities | Ongoing
  To characterize the physiologic, biochemical or genetic basis of theabnormality of immunity.

SECONDARY OUTCOMES:
Assess ability to participate in other studies | ongoing
  To assess the patient's ability to safely tolerate specific aspects of other diagnostic or therapeutic research protocols.
Determine eligibility for other studies | ongoing
  To determine a patient's eligibility for other studies.
Establish baseline of pattern/pace of disease process before participating in therapeutic trials | ongoing
  To establish a baseline assessment of the pace and extent of the disease before entering a therapeutic clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Strober, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaffe JS, Eisenstein E, Sneller MC, Strober W. T-cell abnormalities in common variable immunodeficiency. Pediatr Res. 1993 Jan;33(1 Suppl):S24-7; discussion S27-8. doi: 10.1203/00006450-199305001-00128. PMID 7679486
- [Background] Mannon PJ, Fuss IJ, Dill S, Friend J, Groden C, Hornung R, Yang Z, Yi C, Quezado M, Brown M, Strober W. Excess IL-12 but not IL-23 accompanies the inflammatory bowel disease associated with common variable immunodeficiency. Gastroenterology. 2006 Sep;131(3):748-56. doi: 10.1053/j.gastro.2006.06.022. PMID 16952544
- [Background] Cunningham-Rundles C. Autoimmune manifestations in common variable immunodeficiency. J Clin Immunol. 2008 May;28 Suppl 1(Suppl 1):S42-5. doi: 10.1007/s10875-008-9182-7. Epub 2008 Mar 6. PMID 18322785
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1989-I-0158.html